CLINICAL TRIAL: NCT06636682
Title: A Multicenter, Adaptive, Phase 2, Randomized, Open-label Study of Irradiated Autologous Cellular Vaccine in Men With High-Risk Prostate Cancer Following Prostatectomy
Brief Title: FK-PC101 as Adjuvant Therapy for Men With High-Risk Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cellvax Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FK-PC101-01
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer (Adenocarcinoma); Prostate CA; Prostate Cancers; Prostate Cancer (Post Prostatectomy); Prostate Cancer; Prostate Cancer Patients Undergoing Radical Prostatectomy; High-risk Prostate Cancer
Keywords: Vaccine; Prostatectomy; Autologous; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- FK-PC101 (Experimental): Up to 7 doses of intradermal FK-PC101 vaccine
  Interventions: Biological: FK-PC101
- Standard of Care (Active Comparator): Standard of care, with possibility to cross-over to FK-PC101 vaccine should prostate cancer recur within 1 year of radical prostatectomy
  Interventions: Biological: Standard of Care (SOC)

INTERVENTIONS:
Biological: FK-PC101 — Up to 7 doses of FK-PC101 will be administered intradermally between Day 1 and Day 180. The immune adjuvant Bacillus Calmette Guérin (BCG) will be given concurrently with Dose 1 (day 1) and Dose 2 (day 8).
  Arms: FK-PC101
Biological: Standard of Care (SOC) — Subject receives Investigator-defined standard of care, excluding adjuvant therapy. If prostate cancer recurs before 12 months after radical prostatectomy, subjects are eligible to receive up to 7 doses of intradermal FK-PC101 vaccine (first 2 given concurrently with BCG).
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to learn if the vaccine FK-PC101 works to delay or prevent the return of prostate cancer in men who have had surgery to remove their prostate cancer. It will also learn about the safety of FK-PC101. The main questions it aims to answer are:

Does FK-PC101 delay or prevent the return of prostate cancer following surgery? What medical problems do participants (subjects) have when taking FK-PC101?

Researchers will compare FK-PC101 to current treatment practice to see if FK-PC101 works to prevent or delay the return of prostate cancer following surgery to remove the prostate cancer tumor.

Subjects will:

Have a sample of the prostate cancer tissue collected at the time of surgery to remove this tissue from the body. This tissue will then be used to create a personalized vaccine that is specific to your prostate cancer.

If randomly selected to receive the vaccine, subjects will receive the vaccine up to 7 times over a 6-month period.

In addition to the treatment visits for those randomized to receive FK-PC101, there will be up to 4 follow up visits to the clinic over a 22-month (nearly 2 year) period.

For subjects randomized to receive current treatment practice, they will be asked to attend up to 8 visits over 22 months to track if there is any detectable cancer. Should their prostate cancer return within a year following surgery, they will be eligible to receive FK-PC101, which already had been produced and thus no additional tumor tissue would need to be obtained.

Subjects in both study arms will have regular blood tests and scans to test whether their prostate cancer has returned.

DETAILED DESCRIPTION:
This is a multicenter, adaptive, Phase 2, randomized, open-label study designed to evaluate the efficacy of FK-PC101 adjuvant therapy in men with localized prostate cancer who have undergone radical prostatectomy (RP). Subjects will undergo a 3-step screening and enrollment process. Following an initial safety run-in that will include at least three subjects assigned to receive FK-PC101 vaccine and monitored closely for safety, subjects randomized to the vaccine group will receive up to 7 doses of FK-PC101, starting at 2 months post-RP. Subjects in the control group will receive standard-of-care. All subjects will have assessments at 60 days (2 months), 90 days (3 months) and 180 days (6 months) and then continue with follow-up visits at 10, 14, 18, and 22 months after randomization.

FK-PC101 is an autologous cellular vaccine, with each product being manufactured from a portion of tumor from each subject's prostatectomy specimen. The primary endpoint of DFS will be compared with the control group, who will also meet all eligibility criteria but who do not receive any postoperative adjuvant therapy.

Subjects will undergo a three-step eligibility process with criteria prior to RP, immediately following RP and 2 months post-RP/immediately prior to randomization.

Subjects will be randomized in a 1:1 open-label fashion to the vaccine group and the control group. Subjects will be stratified based on pathologic nodal status (pN0 vs. pN1). Subjects in the vaccine group will initiate vaccine dosing with up to 7 doses given between Day 1 and Day 180 (on Days 1, 8, 15, 22, 60, 90 and 180). Subjects randomized to the control group will be followed through 8 follow-up visits through month 22 (2 years post-surgery).

Following disease recurrence, all subjects may be treated with other prostate cancer therapies as deemed appropriate. Subjects in the control group will be eligible to receive their vaccine after disease recurrence has been documented. For subjects in the control group who elect to receive their vaccine, it must be started within 1 year of randomization. The vaccine doses may be administered prior to, during, or following other prostate cancer therapies but will follow the same schedule as for the subjects in the vaccine group.

ELIGIBILITY:
Inclusion Criteria:

* Has localized high-risk or very high-risk prostate cancer based on the NCCN v4.2023 classification.
* Has ≥3 prostate biopsy cores with ≥50% tumor involvement.
* Has PSA >4 ng/mL ≤28 days prior to enrollment.
* Has no evidence of distant metastases based on PSMA-PET/CT performed ≤28 days prior to enrollment.
* Is a candidate for radical prostatectomy, and scheduled radical prostatectomy date must be 3 to 14 days after enrollment.
* Has not received nor plans to receive neoadjuvant (preoperative) radiation therapy, androgen deprivation therapy (ADT), or any other anticancer therapy.
* Has a life expectancy >5 years.

Additional key eligibility criteria immediately postoperative for inclusion in the randomized population include:

* Stage >pT3a (tumor has extended outside of the prostate on one side).
* Gleason score of 8, 9, or 10 (high/very high) on prostatectomy specimen.
* Subjects with pT3b or pT4 tumors with a Gleason sum 7 (4+3) are eligible.
* Pelvic lymph node dissection (PLND) is required with either pN0 or pN1 nodal staging permitted.
* Subjects must have negative surgical margins or microscopic-only positive surgical margins.

Final eligibility criteria at 2 months postoperative for randomization include:

* FK-PC101 has been produced for the subject and meets all release specifications.
* An undetectable PSA (<0.04 ng/mL) on the most recent test performed prior to randomization (Day -4 to -7).
* No prior, current, or planned future postoperative or adjuvant XRT, hormonal therapy such as ADT, or any other anticancer therapy (future therapy should not be administered until evidence exists of prostate cancer disease recurrence [such as PSA recurrence]).
* Adequate organ function based on CBC and chemistry studies within 2 weeks of Day 1 (Day -14 to -7). Specific laboratory requirements include:

  * Absolute neutrophil count (ANC) >1000/µL
  * Platelet count >100,000/µL.
  * Hemoglobin >8.0 gm/dL.
  * Estimated glomerular filtration rate (eGFR) >60 mL/minute based on Cockcroft-Gault formula.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both <2 × upper limit of normal (ULN).
  * Albumin >3.0 gm/dL.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions of the study.

Exclusion Criteria:

* Has an additional active malignancy that may confound the assessment of the study endpoints. If the subject has a past cancer history (active malignancy within 2 years prior to study entry) with substantial potential for recurrence, this must be discussed with the Sponsor before study entry. Note: Subjects with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer and carcinomas in situ (including breast DCIS, transitional cell carcinoma/NMIBC, anal carcinoma, and melanoma in situ).
* Is eligible for and elects to receive adjuvant therapy following RP.
* Has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association [NYHA] Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina, pulmonary embolism or stroke within 6 months prior to study entry, uncontrolled hypertension, or clinically significant arrhythmias not controlled by medication).
* Has uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the subject at significant risk for pulmonary complications during the study.
* Has known metastases, such as bone, visceral, or brain or leptomeningeal metastases.
* Has an active autoimmune disease or Grade ≥3 pneumonitis that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) or treatment with drugs (e.g., neomercazol, carbamazole) that function to decrease the generation of thyroid hormone by a hyperfunctioning thyroid gland (e.g., in Graves' disease) is not considered a form of systemic treatment of an autoimmune disease.
* Is currently receiving systemic steroid therapy at a prednisone equivalent dose of >10 mg daily for at least 1 week or other form of immunosuppressive therapy within 7 days prior to enrollment.
* Has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
* Is at risk for disseminated BCG infection or has previously demonstrated an allergic response to BCG or its components.
* Has known positive status for human immunodeficiency virus (HIV) or active or chronic Hepatitis (Hep) B or Hep C. Screening is not required.
* Has any medical condition which in the opinion of the Investigator places the subject at an unacceptably high risk for toxicity.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-05-04 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Up to approximately 22 months
  DFS is defined as local prostate cancer recurrence, distant metastatic prostate cancer recurrence, biochemical recurrence of PSA, or death from any cause

SECONDARY OUTCOMES:
Time to next treatment (TTNT) | Up to approximately 22 months
  Time from randomization until disease recurrence or receipt of any form of adjuvant or salvage radiotherapy, hormonal therapy including ADT, or any other form of prostate cancer therapy post-randomization
Metastasis-free survival (MFS) | Up to approximately 22 months
  Time from date of randomization to the 1st evidence of distant metastatic prostate cancer recurrence as detected by PSMA-PET/CT or other imaging performed, or to death from any cause
Immune response to FK-PC101 | From baseline until Month 22
  Immune response to FK-PC101 as measured by ELISpot assay (FK-PC101 arm only)
Safety and tolerability of FK-PC101 | Up to approximately 22 months
  Frequency and severity of AEs per the NCI-CTCAE version 5.0

OTHER OUTCOMES:
Overall survival (OS) | Up to approximately 22 months
  Time from date of randomization to date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Kreutz, MD PhD, Study Chair — Cellvax Therapeutics Inc
Locations (3):
- United States (3):
  - University of Chicago Medicine, High-Risk and Advanced Prostate Cancer Clinic, Chicago, Illinois
  - Central Ohio Urology Group, Gahanna, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No